CLINICAL TRIAL: NCT01345773
Title: Incidence of Venous Thromboembolism Following Surgery in Patients With Gastric Cancer; a Prospective Study
Brief Title: Incidence of Venous Thromboembolism Following Surgery in Patients With Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Keun-Wook Lee, M.D. & Ph.D., Seoul National University Bundang Hospital
Other Study IDs: GC-VTE-01
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Gastric Cancer; Venous Thromboembolism; Postoperative Period
MeSH Terms: conditions — Stomach Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving gastric cancer surgery
  Interventions: Procedure: Gastric surgery

INTERVENTIONS:
Procedure: Gastric surgery — Patients receiving gastric cancer surgery will be prospectively observed for the development of venous thromboembolism

SUMMARY:
Venous thromboembolism (VTE) has considerably harmful effects on morbidity and mortality of cancer patients. Several guidelines recommendations have been made about the use of anticoagulation for the prevention and treatment of VTE in Western patients with cancer. In Western VTE guidelines, all solid cancer patients receiving abdominal major surgery are strongly recommended to receive pharmacologic prophylactic anticoagulation such as low molecular weight heparin (LMWH) in the perioperative periods. These guideline recommendations are based on high incidence of postoperative VTE development in Western cancer patients. However, there have been many cumulative data about the effect of different ethnicity on the VTE development and more and more investigators and clinicians admit that Asian ethnicity has lower incidence of VTE than Western ethnicity. Therefore, it may not be advisable to apply Western guidelines as it is to the clinical situation of Asian cancer patients.

Although gastric cancer is the common cancer in Asia, there is no prospective data on the incidence of VTE development during the postoperative period of gastric cancer surgery. In other words, Asian doctors including Korean clinicians don't know the exact incidence of surgery-related VTE. From their clinical experiences, most Korean surgeons think that the incidence of postoperative VTE development is rare. They also have much concern about the complications such as bleeding that might be caused by routine use of pharmacologic thromboprophylaxis during the perioperative periods. Therefore, in most clinical situation, Korean surgeons do not perform perioperative pharmacologic thromboprophylaxis using LMHW. Considering these clinical situations in Korea, the uncritical acceptance of Western guidelines is inappropriate. The necessity of pharmacologic thrombo-prophylaxis can be answered only from the results of the prospective study on the incidence of postoperative VTE development after gastric cancer surgery. Moreover, current surgical trend in cancer patients is minimally invasive approach such as laparoscopic surgery. However, the necessity of pharmacologic thromboprophylaxis in patients receiving laparoscopic cancer surgery has not been evaluated even in Western countries. Western guidelines also cannot exactly answer whether pharmacologic thromboprophylaxis is really necessary in cancer patients receiving laparoscopic cancer surgery. On above backgrounds, this study was designed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of stomach or gastroesophageal junction
* Age ≥ 20 years
* Patients receiving curative or palliative abdominal surgery (lasting ≥ 30 minutes) (both open and laparoscopic surgery will be included)

Exclusion Criteria:

* No histological confirmation
* Patients who already have VTE (or pulmonary embolism) at the screening periods of this study
* Past medical history of VTE or pulmonary embolism
* Patients with the history of other cancer (Patients who were disease-free for > 5 years from previous other cancer is allowed to be included in this study)
* Patients with thrombophilia or other comorbidities requiring anticoagulation (i.e. atrial fibrillation or cerebral infarct requiring anticoagulation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer receiving curative or palliative gastric cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The incidence of symptomatic or asymptomatic VTE | 5~12 days after the gastric cancer surgery (by doppler US) or the follow-up period of postoperative 1 month
  To evaluate the incidence of symptomatic or asymptomatic VTE detected by Doppler venous ultrasound during postoperative periods in patients with gastric cancer receiving surgery

SECONDARY OUTCOMES:
Risk factors for the development of VTE | 5~12 days after the gastric cancer surgery (by doppler US) or the follow-up period of postoperative 1 month
  To identify risk factors for the development of VTE in this population

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea